CLINICAL TRIAL: NCT02969564
Title: 18F-NaF-PET/MR vs 99mTc-MDP-SPECT/CT to Detect Bone Metastases in Prostate Cancer Patients.
Status: Completed | Type: Observational
Sponsor: Valentina Garibotto (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor-Investigator, Valentina Garibotto, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 15-118
Record Dates: First submitted 2016-04-21; First posted 2016-11-21 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Bone Metastases; Prostate Cancer
Keywords: prostate cancer; bone metastases; PET/MRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- prostate cancer patient, with up to five metastases: prostate cancer patient, with up to five metastases (oligo-bone metastatic) based on scintigraphy 99mTc-MDP-SPECT/CT.
  Interventions: Other: scintigraphy 99mTc-MDP-SPECT/CT.; Other: 18F-NaF-PET/MR

INTERVENTIONS:
Other: scintigraphy 99mTc-MDP-SPECT/CT. — SPECT/CT will be performed for every patient in the frame of their clinical follow up
Other: 18F-NaF-PET/MR — a 18F-NaF-PET/MR will be performed, in the frame of this clinical study, to the patients to assess the difference of sensitivity of the 2 exams

SUMMARY:
The number of metastases in a patient with primary or recurrent prostate cancer has major prognostic implication.

The purpose is to compare, in a pilot study, the diagnostic performance of 18F-NaF-PET/MR with respect to the results of the scintigraphy 99mTc-MDP-SPECT/CT (routine exam) for determining the presence or absence of bone lesions in prostate cancer patient, with up to five metastases (oligo-bone metastatic) based on scintigraphy 99mTc-MDP-SPECT/CT. The gold standard will be a combination of clinical follow-up, additional imaging and biopsy, as indicated by the multidisciplinary discussion at the tumor board. The findings from whole-body 99mTc-MDP-SPECT/CT, 18F-NaF-PET/MR, and the combination of the 2 modalities will be categorized by 2 teams of 2 readers as benign or probably benign, equivocal, or malignant or probably malignant and compared with the results of follow-up for JAFROC and ROC analysis.

ELIGIBILITY:
Inclusion Criteria:

* Oligo- metastatic patient with prostate cancer and bone lesions (up to five metastases) based on scintigraphy and whole-body SPECT/CT (staging or recurrence).
* Patient must be able to provide informed consent.
* Patient is ≥ 18 years old

Exclusion Criteria:

* Patient with another active malignancy.
* Patient is < 18 years old
* Patients with contraindications of MRI procedure (metal implants, cardiac pacemakers, old type of prosthesis)
* Patients with severe renal impairment (MDRD < 30)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oligo- metastatic patient with prostate cancer and bone lesions (up to five metastases)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Compare the diagnostic performance of 18F-NaF-PET/MR scanning to that of whole body 99mTc-MDP-SPECT/CT for detecting cancer that has spread to the bone (bone metastasis) | through study completion, an average of 2 years
  the primary measure will be differences in the area under the curves (AUC) of the receiver operating characteristic (ROC) curves that will be generated from the interpretations of each technology.

SECONDARY OUTCOMES:
To assess differences in sensitivity and specificity in detecting bone metastases between the two imaging modalities. | through study completion, an average of 2 years
  Sensitivity and specificity of PET and SPECT for the detection of secondary bone lesions (gold standard: clinical and imaging follow up)
To determine the number of equivocal and diagnostic tests resulting from the two imaging modalities. | through study completion, an average of 2 years
  rate of equivocal/non equivocal findings for the two modalities

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospital, Geneva, Switzerland